CLINICAL TRIAL: NCT01020227
Title: A Randomized Controlled Trial to Assess the Usefulness of Integrative Medicine Tools As Adjunctive Care for Women After Coronary Artery Bypass Grafting
Brief Title: Usefulness of Integrative Medicine Tools As Adjunctive Care for Women After Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Erin L Olivo PhD, MPH, Assistant Clinical Professor of Medical Psychology ( In Psychiatry), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAB1732
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Disease
Keywords: Postoperative Care; Quality of Life; Integrative Medicine; Coronary Artery Bypass Graft Surgery
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrative Therapies (Experimental): Patients in the intervention group were given a cardiac yoga video, a guided imagery audiotape, instruction in diaphragmatic breathing, and an educational booklet outlining recommendations for dietary change. Patients were followed for 6 months by a health educator who provided ongoing education and encouragement
  Interventions: Behavioral: Integrative Therapies Intervention
- Standard Care (No Intervention): Patients were given no intervention but were contacted at 6 weeks and 6 months for data collection purposes

INTERVENTIONS:
Behavioral: Integrative Therapies Intervention — Patients in the intervention group were given a cardiac yoga video, a guided imagery audiotape, instruction in diaphragmatic breathing, and an educational booklet outlining recommendations for dietary change. Patients were followed for 6 months by a health educator who provided ongoing education and encouragement
  Arms: Integrative Therapies

SUMMARY:
Background: This randomized controlled trial investigates the effectiveness of an Integrative Therapies (IT) health education intervention in improving physical and psychological functioning in female patients after coronary artery bypass graft (CABG).

Methods: One hundred female cardiac surgery patients were assigned to either an intervention or standard care control group. Patients in the intervention group were given a cardiac yoga video, a guided imagery audiotape, instruction in diaphragmatic breathing, and an educational booklet outlining recommendations for dietary change. Patients were followed for 6 months by a health educator who provided ongoing education and encouragement and were assessed at 6 weeks and 6 months post surgery to determine between group differences on physical functioning and psychological distress using the SF-36 and the Profile of Mood States

DETAILED DESCRIPTION:
Coronary artery disease is the most frequent cause of death for women in the United States. Increasingly coronary artery bypass graft (CABG) surgery is used for women as a treatment for this disease and women now account for nearly 30% of patients undergoing CABG surgery. Women are reported to have higher morbidity and mortality after CABG surgery than men. In addition to this higher complication and death rate, recent studies suggest that women experience more fear, stress, depression and anxiety before and after surgery than men. This randomized, controlled study was developed to research the feasibility and possible effects of providing health education and complementary and alternative medicine (CAM) tools to women after they have undergone cardiac surgery.

This study is a randomized controlled clinical trial of 150 women from the Columbia campus of New York Presbyterian Hospital who recently had cardiac surgery. Baseline information on risk factor status, psychosocial status, quality of life, and CAM usage and expectancy will be obtained on all participants. Women will be randomized to CAM health education or standard care and will be followed for 6 months. Patients randomized to CAM health education will receive a three-tiered program in CAM education by a certified or trained practitioner in Yoga, Guided Imagery, and Nutrition. Patients will receive both personalized instruction in use of these CAM therapies and custom-designed instructional material including a:

1. videotape on cardiac yoga,
2. a guided imagery audiotape and
3. a booklet on micronutritional approaches to cardiac care (developed by Dr Oz and the Columbia Integrative Medicine Program)

Women randomized to CAM health education will be contacted at 2, 4, and 6 weeks, 3 months, and 6 months post surgery to assess progress toward reaching prevention goals, their utilization of CAM therapies, and their impact on psychological and physical health. The health educator will problem solve with the patient to overcome barriers toward reaching prevention and CAM goals.

Assessments of the following outcomes will be made at 6 weeks and 6 months post intervention: overall mood as measured by the Profile of Mood States12, perception of stress as measured by a single-item, likert stress scale, psychological and mental health status as measured by the SF36, and the occurrence of major adverse cardiac events (cardiovascular disease death, nonfatal myocardial infarction, myocardial revascularization procedure, stroke, non-coronary arterial revascularization, cardiovascular hospitalizations).

It is hypothesized that the CAM education intervention is a feasible mode of disseminating information and encouraging the use of CAM tools to women post cardiac surgery. It is also hypothesized that the CAM intervention will increase overall mood (POMS), will decrease perceived stress (self report stress score), will increase self report of physical and mental functioning (SF36, PH and MH scales) and will decrease episodes of major adverse cardiac events at 6 months postsurgery.

Data analysis will include evaluation of the following within group outcomes: overall adherence and utilization of CAM tools, overall frequency of use by tool (yoga, guided imagery, dietary changes), time point of initiation of CAM use, frequency of use by demographics (age, ethnicity, surgery type, previous CAM exposure, employment status, marital status), most frequent barriers to use, rate of refusal, rate of dropout. In addition, comparisons of the between group outcomes (Mood, Stress, and Physical and Mental Functioning) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Undergoing CABG or Valve Surgery

Exclusion Criteria:

* Non-English speaking
* No home phone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Self reported psychosocial adjustment | 6 weeks and 6 months post surgery

SECONDARY OUTCOMES:
Self reported physical functioning and clinical cardiovascular outcomes | 6 weeks and 6 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Olivo, PhD, MPH, Principal Investigator — Columbia University; Mehmet C Oz, MD, Study Chair — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States